CLINICAL TRIAL: NCT06410209
Title: Walking Juntos: Developing and Testing a Culturally-Tailored Mobile Health and Social Media Physical Activity Intervention Among Adolescent and Young Adult Childhood Cancer Survivors
Brief Title: A Culturally-Tailored Mobile Health and Social Media Physical Activity Intervention for Improving Physical Activity in Hispanic or Latino/Latina Adolescent and Young Adult Childhood Cancer Survivors, Walking Juntos Study
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Children's Oncology Group (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Triple | Purpose: Prevention
Other Study IDs: ALTE2321; NCI-2024-03609 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); ALTE2321 (Other: Children's Oncology Group); COG-ALTE2321 (Other: DCP); ALTE2321 (Other: CTEP); R01CA274450 (NIH); UG1CA189955 (NIH)
Record Dates: First submitted 2024-05-07; First posted 2024-05-13 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: Hematopoietic and Lymphatic System Neoplasm; Malignant Solid Neoplasm
MeSH Terms: interventions — Organizational Objectives; Interviews as Topic

STUDY DESIGN:
Who Masked: Care Provider, Investigator, Outcomes Assessor
Masking Description: Investigators and participating site staff are blinded.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Stage 1 (Fitbit, interview) (Experimental): Patients wear a Fitbit physical activity tracker daily, set physical activity goals, receive text messages, and view private social media peer support group content over 7-10 days once every 3 months. Patients also wear a research grade activity measuring device over 1-3 days and participate in a one-on-one interview once every 3 months for 9 months. (COMPLETE 10/30/2025)
  Interventions: Other: Goal Setting; Other: Interview; Other: Media Intervention; Other: Medical Device Usage and Evaluation; Other: Questionnaire Administration; Other: Text Message-Based Navigation Intervention
- Stage 2, Group I (Fitbit, goal setting, peer support) (Experimental): INTENSIVE PHASE: Patients wear a Fitbit physical activity tracker daily and receive weekly reminders to wear the Fitbit for 12 weeks. Patients attend weekly goal setting sessions, receive individualized physical activity goals, view and post private social media peer support group content 2-3 times weekly, receive badges, and participate in a monthly Zoom meeting with their peers to discuss physical activity for 12 weeks. Patients may optionally choose a physical activity partner. Partners wear a Fitbit physical activity tracker and receive educational materials about supporting the participant.
  MAINTENANCE PHASE: Patients wear a Fitbit physical activity tracker daily and set their own physical activity goals weekly for 4 weeks. Patients also receive access to the social media account and post content for 4 weeks. In addition, patients may continue to have their physical activity partner support them as in the Intensive Phase.
  Interventions: Other: Discussion; Other: Goal Setting; Other: Interview; Other: Media Intervention; Other: Medical Device Usage and Evaluation; Other: Questionnaire Administration; Other: Reward; Other: Text Message-Based Navigation Intervention
- Stage 2, Group II (Fitbit) (Active Comparator): Patients wear a Fitbit physical activity tracker daily for 12 weeks.
  Interventions: Other: Medical Device Usage and Evaluation; Other: Questionnaire Administration

INTERVENTIONS:
Other: Discussion — Participate in Zoom meetings with peers to discuss physical activity
  Other Names: Discuss
  Arms: Stage 2, Group I (Fitbit, goal setting, peer support)
Other: Goal Setting — Set physical activity goals
  Arms: Stage 1 (Fitbit, interview); Stage 2, Group I (Fitbit, goal setting, peer support)
Other: Interview — Participate in a one-on-one interview
  Arms: Stage 1 (Fitbit, interview)
Other: Interview — Ancillary studies
  Arms: Stage 2, Group I (Fitbit, goal setting, peer support)
Other: Media Intervention — View private social media peer support group content
  Arms: Stage 1 (Fitbit, interview); Stage 2, Group I (Fitbit, goal setting, peer support)
Other: Medical Device Usage and Evaluation — Wear a Fitbit physical activity tracker
Other: Medical Device Usage and Evaluation — Wear a research grade activity measuring device
  Arms: Stage 1 (Fitbit, interview)
Other: Questionnaire Administration — Ancillary studies
Other: Reward — Receive badges
  Arms: Stage 2, Group I (Fitbit, goal setting, peer support)
Other: Text Message-Based Navigation Intervention — Receive text messages
  Other Names: Automated Text Message-Based Navigation; Text Message-Based Navigation
  Arms: Stage 1 (Fitbit, interview)
Other: Text Message-Based Navigation Intervention — Receive reminders
  Other Names: Automated Text Message-Based Navigation; Text Message-Based Navigation
  Arms: Stage 2, Group I (Fitbit, goal setting, peer support)

SUMMARY:
This clinical trial tests the impact of a culturally-tailored home-based physical activity program on physical fitness in Hispanic or Latino/Latina adolescent and young adult (AYA) childhood cancer survivors. After treatment for cancer, some AYA survivors experience long-term effects from the cancer and its treatment including weight gain, fatigue and decreased physical fitness. Hispanic or Latino/Latina survivors may have a higher risk of these effects compared to non-Hispanics. Regular physical activity helps maintain healthy weight, energy levels and overall health. Participating in a culturally-tailored home-based physical activity program may help increase physical activity in Hispanic or Latino/Latina AYA childhood cancer survivors.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Use an iterative approach to develop a culturally-tailored multilevel remote-based physical activity (PA) intervention among a total of 20 Latinx adolescent and young adult survivors of childhood cancer (AYA survivors), 8-12 whose preferred language is English and 8-12 whose preferred language is Spanish, using the StepByStep intervention as a starting point. (Stage 1) II. Conduct a randomized controlled trial (RCT) to test the potential efficacy of the culturally-tailored remote-based PA intervention (versus [vs.] Fitbit PA tracker only) with respect to the primary outcome of moderate to vigorous physical activity (MVPA) measured with a validated, wearable Fitbit PA tracker over 12 weeks among a separate group of 170 Latinx AYA survivors whose preferred language is Spanish or English (n=85 per randomization group) and who do not meet PA guidelines at timepoint (T) 1. The control group will receive a Fitbit only. (Stage 2)

SECONDARY OBJECTIVES:

I. Among the patients enrolled to the RCT component of the study, evaluate the potential efficacy of randomization to the intervention group relative to control group with respect to decreasing sedentary time as assessed by a Fitbit PA tracker.

II. Evaluate potential efficacy of randomization to the active intervention group with respect to improvement in reported health-related quality of life.

EXPLORATORY OBJECTIVES:

I. Evaluate potential efficacy of randomization to the active intervention group with respect to physiological measurements predictive of cardiometabolic health.

II. Determine the acceptability of and guidance on improving the intervention phases in preparation for a fully powered, long term RCT by conducting two rounds of post-trial qualitative interviews among participants in the intervention Group n=12-15 for the intensive intervention phase and n=12-15 for the maintenance intervention phase. Preferences and barriers for an additional diet and nutrition component will also be explored.

OUTLINE:

STAGE 1: Patients wear a Fitbit physical activity tracker daily, set physical activity goals, receive text messages, and view private social media peer support group content over 7-10 days once every 3 months. Patients also wear a research grade activity measuring device over 1-3 days and participate in a one-on-one interview once every 3 months for 9 months.

STAGE 2: Patients are randomized to 1 of 2 groups.

GROUP I (INTERVENTION):

INTENSIVE PHASE: Patients wear a Fitbit physical activity tracker daily and receive weekly reminders to wear the Fitbit for 12 weeks. Patients attend weekly goal setting sessions, receive individualized physical activity goals, view and post private social media peer support group content 2-3 times weekly, receive badges, and participate in a monthly Zoom meeting with their peers to discuss physical activity for 12 weeks. Patients may optionally choose a physical activity partner. Partners wear a Fitbit physical activity tracker and receive educational materials about supporting the participant.

MAINTENANCE PHASE: Patients wear a Fitbit physical activity tracker daily and set their own physical activity goals weekly for 4 weeks. Patients also receive access to the social media account and post content for 4 weeks. In addition, patients may continue to have their physical activity partner support them as in the Intensive Phase.

GROUP II (CONTROL): Patients wear a Fitbit physical activity tracker daily for 12 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Patient must be ≥ 15 years and < 21 years at the time of enrollment
* First diagnosis of malignant neoplasm (International Classification of Diseases for Oncology [ICD-O] behavior code of "3") in first and continuous remission at the time of enrollment
* Curative cancer treatment must have included chemotherapy (including cellular therapy) and/or radiation (including radioactive iodine). Note: Certain stem cell transplant procedures are excluded. Reminder: Children's Oncology Group (COG) therapeutic trial participation is not required
* Completed all chemotherapy and/or radiation therapy in the last 3-36 months. This includes completion of all oral (e.g., tyrosine kinase inhibitors) and/or maintenance chemotherapy
* Self-report of < 420 minutes of moderate-to-vigorous physical activity per week as assessed and documented via the study-specific Physical Activity Worksheet. Note: See the case report forms packet on the COG study web page for the study specific Physical Activity Worksheet
* Ambulatory and no known medical contraindications to increasing physical activity
* No known significant physical or cognitive impairment that would prevent use of the electronic devices used for the protocol intervention (e.g., Fitbit, smartphone, tablet, or computer)
* Able to read and write Spanish or English
* Self-identify as Hispanic, Latino/Latina/Latinx

Exclusion Criteria:

* Patients with previous allogeneic hematopoietic stem cell transplant (HSCT) are excluded. Note: Patients with previous autologous HSCT, chimeric antigen receptor T-cell (CAR T-cell) therapy, and other cellular cancer therapies can participate as long as all other eligibility criteria are satisfied
* Post-menarchal female patients who are pregnant or planning to become pregnant in the next year are excluded. Note: Pregnancy status can be established by clinical history with patient. Post-menarchal female patients are eligible as long as they agree to use an effective contraceptive method (including abstinence) during study participation
* Participants who were enrolled in ALTE2031 (Step by Step) cannot enroll in ALTE2321. Participants who were enrolled in ALTE2321 stage 1 (cultural tailoring) cannot enroll to participate in stage 2 (RCT)
* All patients and/or their parents or legal guardians must sign a written informed consent. Note: Informed consent may be obtained electronically/online if allowed by local site policy and institutional review board (IRB)/research ethics board (REB) of record
* All institutional, Food and Drug Administration (FDA), and National Cancer Institute (NCI) requirements for human studies must be met

Ages: 15 Years to 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 190 (Estimated)
Dates: Start 2024-10-15 (Actual); Primary Completion 2027-09-15 (Estimated); Study Completion 2027-09-15 (Estimated)

PRIMARY OUTCOMES:
Moderate to vigorous physical activity (MVPA) | Baseline to 11-12 weeks post randomization
  MVPA will be measured by active minutes using Fitbit. Will report the mean change from baseline to the 11-12-week post randomization timepoint by trial arm alongside corresponding confidence intervals estimated under a linear mixed effects model.

SECONDARY OUTCOMES:
Sedentary time | Baseline to 11-12 weeks post randomization
  Sedentary time as measured by FitBit. Will report the mean change from baseline to the 11-12-week post randomization timepoint by trial arm alongside corresponding confidence intervals estimated under a linear mixed effects model.
Global functioning | Baseline to 11-12 weeks post randomization
  Global functioning will be measured using Spanish language versions of the Pediatric Quality of Life inventory (PedsQL) 4.0 Generic Core Scales. Will report the mean change from baseline to the 11-12-week post randomization timepoint by trial arm alongside corresponding confidence intervals estimated under a linear mixed effects model.
Physical functioning | Baseline to 11-12 weeks post randomization
  Physical functioning will be measured using Spanish language versions of the PedsQL 4.0 Generic Core Scales. Will report the mean change from baseline to the 11-12-week post randomization timepoint by trial arm alongside corresponding confidence intervals estimated under a linear mixed effects model.
Social functioning | Baseline to 11-12 weeks post randomization
  Social functioning will be measured using Spanish language versions of the PedsQL 4.0 Generic Core Scales. Will report the mean change from baseline to the 11-12-week post randomization timepoint by trial arm alongside corresponding confidence intervals estimated under a linear mixed effects model.
Fatigue | Baseline to 11-12 weeks post randomization
  Fatigue will be measured using the18-item PedsQL 4.0 Multidimensional Fatigue Scale in Spanish or English. Will report the mean change from baseline to the 11-12-week post randomization timepoint by trial arm alongside corresponding confidence intervals estimated under a linear mixed effects model.

OTHER OUTCOMES:
Change in cardiopulmonary fitness | At baseline and up to final evaluation at 11-12 weeks post-randomization
  Change in cardiopulmonary fitness will be assessed by Fitbit cardio fitness score and heart rate.
Change in resting heart rate | At baseline and up to final evaluation at 11-12 weeks post-randomization
  Change in resting heart rate will be measured by Fitbit cardio fitness score and heart rate.

CONTACTS AND LOCATIONS:
Overall Officials: Jason A Mendoza, Principal Investigator — Children's Oncology Group
Locations (77):
- United States (76):
  - Banner Children's at Desert, Mesa, Arizona
  - Phoenix Childrens Hospital, Phoenix, Arizona
  - Arkansas Children's Hospital, Little Rock, Arkansas
  - Kaiser Permanente Downey Medical Center, Downey, California
  - City of Hope Comprehensive Cancer Center, Duarte, California
  - Miller Children's and Women's Hospital Long Beach, Long Beach, California
  - Mattel Children's Hospital UCLA, Los Angeles, California
  - Valley Children's Hospital, Madera, California
  - UCSF Benioff Children's Hospital Oakland, Oakland, California
  - Kaiser Permanente-Oakland, Oakland, California
  - Rady Children's Hospital - San Diego, San Diego, California
  - Children's Hospital Colorado, Aurora, Colorado
  - Yale University, New Haven, Connecticut
  - Alfred I duPont Hospital for Children, Wilmington, Delaware
  - MedStar Georgetown University Hospital, Washington D.C., District of Columbia
  - Golisano Children's Hospital of Southwest Florida, Fort Myers, Florida
  - Memorial Regional Hospital/Joe DiMaggio Children's Hospital, Hollywood, Florida
  - Nemours Children's Clinic-Jacksonville, Jacksonville, Florida
  - University of Miami Miller School of Medicine-Sylvester Cancer Center, Miami, Florida
  - Miami Cancer Institute, Miami, Florida
  - AdventHealth Orlando, Orlando, Florida
  - Arnold Palmer Hospital for Children, Orlando, Florida
  - Nemours Children's Hospital, Orlando, Florida
  - Nemours Children's Clinic - Pensacola, Pensacola, Florida
  - Johns Hopkins All Children's Hospital, St. Petersburg, Florida
  - Saint Joseph's Hospital/Children's Hospital-Tampa, Tampa, Florida
  - Children's Healthcare of Atlanta - Arthur M Blank Hospital, Atlanta, Georgia
  - Memorial Health University Medical Center, Savannah, Georgia
  - Lurie Children's Hospital-Chicago, Chicago, Illinois
  - University of Illinois, Chicago, Illinois
  - Southern Illinois University School of Medicine, Springfield, Illinois
  - Riley Hospital for Children, Indianapolis, Indiana
  - Ascension Saint Vincent Indianapolis Hospital, Indianapolis, Indiana
  - Blank Children's Hospital, Des Moines, Iowa
  - University of Kentucky/Markey Cancer Center, Lexington, Kentucky
  - Children's Hospital New Orleans, New Orleans, Louisiana
  - Ochsner Medical Center Jefferson, New Orleans, Louisiana
  - Sinai Hospital of Baltimore, Baltimore, Maryland
  - Walter Reed National Military Medical Center, Bethesda, Maryland
  - Children's Hospitals and Clinics of Minnesota - Minneapolis, Minneapolis, Minnesota
  - Children's Hospital and Medical Center of Omaha, Omaha, Nebraska
  - University of Nebraska Medical Center, Omaha, Nebraska
  - University Medical Center of Southern Nevada, Las Vegas, Nevada
  - Sunrise Hospital and Medical Center, Las Vegas, Nevada
  - Alliance for Childhood Diseases/Cure 4 the Kids Foundation, Las Vegas, Nevada
  - Summerlin Hospital Medical Center, Las Vegas, Nevada
  - Renown Regional Medical Center, Reno, Nevada
  - Hackensack University Medical Center, Hackensack, New Jersey
  - Saint Peter's University Hospital, New Brunswick, New Jersey
  - University of New Mexico Cancer Center, Albuquerque, New Mexico
  - Maimonides Medical Center, Brooklyn, New York
  - Montefiore Medical Center - Moses Campus, The Bronx, New York
  - Duke University Medical Center, Durham, North Carolina
  - Wake Forest University Health Sciences, Winston-Salem, North Carolina
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Legacy Emanuel Children's Hospital, Portland, Oregon
  - Penn State Children's Hospital, Hershey, Pennsylvania
  - Saint Christopher's Hospital for Children, Philadelphia, Pennsylvania
  - BI-LO Charities Children's Cancer Center, Greenville, South Carolina
  - East Tennessee Childrens Hospital, Knoxville, Tennessee
  - Saint Jude Children's Research Hospital, Memphis, Tennessee
  - The Children's Hospital at TriStar Centennial, Nashville, Tennessee
  - Dell Children's Medical Center of Central Texas, Austin, Texas
  - Driscoll Children's Hospital, Corpus Christi, Texas
  - Medical City Dallas Hospital, Dallas, Texas
  - UT Southwestern/Simmons Cancer Center-Dallas, Dallas, Texas
  - El Paso Children's Hospital, El Paso, Texas
  - Cook Children's Medical Center, Fort Worth, Texas
  - Baylor College of Medicine/Dan L Duncan Comprehensive Cancer Center, Houston, Texas
  - M D Anderson Cancer Center, Houston, Texas
  - Children's Hospital of San Antonio, San Antonio, Texas
  - Methodist Children's Hospital of South Texas, San Antonio, Texas
  - University of Texas Health Science Center at San Antonio, San Antonio, Texas
  - Seattle Children's Hospital, Seattle, Washington
  - Providence Sacred Heart Medical Center and Children's Hospital, Spokane, Washington
  - Children's Hospital of Wisconsin, Milwaukee, Wisconsin
- University Pediatric Hospital, San Juan, Puerto Rico